CLINICAL TRIAL: NCT05428722
Title: The Effect of Deep Breathing Exercise With Incentive Spirometer Started in the Preoperative Period in Patients Undergoing Open Cardiac Surgery on Pulmonary Function and Complications: A Randomized Controlled Study
Brief Title: Deep Breathing Exercise With Incentive Spirometer Started in the Preoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice ÖNER CENGİZ, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OnerCengizH
Record Dates: First submitted 2022-06-08; First posted 2022-06-23 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Breathing Exercises
Keywords: Cardiac Surgical Procedures; Breathing Exercises; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: randomized conrolled trial in the parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep breathing group (Experimental): The intervention group is the group in which the investigators applied deep breathing exercises with incentive spirometer starting from the preoperative period.
  Interventions: Behavioral: deep breathing exercises with a incentive spirometer
- Control group (No Intervention): The control group is the group that receives standard clinical care.

INTERVENTIONS:
Behavioral: deep breathing exercises with a incentive spirometer — Deep breathing exercise will be explained to the patients with an incentive spirometer (IS), it will be demonstrated in practice and it will be applied from the first day of hospitalization in addition to routine treatment and care. The patient will be informed about whether they are doing it right and their questions will be answered. It will be ensured that the patients start after breakfast in the morning and make 5-10 inspirations, hold her/his breath for 3 seconds and 5-10 expirations per hour with IS until they fall asleep. The research nurse will warn the patients that they should do the exercise every hour, and the alarms of the patients' mobile phones will be set to ring every hour to be a warning. The start and end time of the exercise will be decided together with the patient, and usually the time of waking and going to bed will be taken into account.
  Arms: deep breathing group

SUMMARY:
Open cardiac surgery is an important treatment method that is frequently used in the treatment of complicated atherosclerotic ischemic heart disease and heart valve diseases.

It is emphasized that respiratory functions decrease significantly after cardiac surgery, especially in the immediate post-operative period. Therefore, despite significant progress in the field of cardiopulmonary bypass and anesthesia technique, pulmonary complications after cardiac surgery are still seen as the main cause of other negative outcomes such as morbidity, mortality, and long-term hospitalization.

Cardiac surgery patients are especially at high risk for the development of postoperative pulmonary complications (PPC).

It has been reported that deep breathing exercises improve postoperative lung expansion and ventilation, resulting in a significant reduction in pulmonary complications.

Postoperative respiratory physiotherapy techniques include techniques such as early mobilization, positioning, breathing exercises, active breathing techniques cycle, as well as the use of different mechanical devices such as incentive spirometry (IS), positive expiratory pressure mask therapy, and continuous positive airway pressure. Incentive spirometry (IS) is a mechanical breathing device that provides slow deep breathing and gives visual feedback and is used as one of the important interventions in the prevention of PPC in patients who have been undergoing open heart surgery for many years.

In studies examining the effectiveness of deep breathing exercise with IS on the development of PPC in open cardiac surgery patients, it is seen that IS application is performed in the postoperative period , it is noteworthy that there is no study examining the effectiveness of preoperative IS application. In the light of this information, the aim of this study is to evaluate the effect of deep breathing exercise with incentive spirometry initiated in the preoperative period on pulmonary function and complications in patients undergoing open heart surgery.

DETAILED DESCRIPTION:
Open cardiac surgery is an important treatment method that is frequently used in the treatment of complicated atherosclerotic ischemic heart disease and heart valve diseases. Complications after cardiac surgery include; supraventricular tachycardia, atrial fibrillation, bradycardia, perioperative myocardial infarction, cardiac arrest, Postoperative pulmonary complications (PPC) such as pneumonia, atelectasis and pleural effusion . It is emphasized that respiratory functions decrease significantly after cardiac surgery, especially in the immediate post-operative period. Therefore, despite significant progress in the field of cardiopulmonary bypass and anesthesia technique, pulmonary complications after cardiac surgery are still seen as the main cause of other negative outcomes such as morbidity, mortality, and long-term hospitalization. Cardiac surgery patients are especially at high risk for the development of PPC. In approximately one-quarter of patients who undergo cardiac surgery without chronic respiratory dysfunction, a mild respiratory tract infection develops ranging from oxygen therapy to acute respiratory failure requiring invasive or non-invasive mechanical ventilation support. Among the factors that cause the development of PPC; surgical stress and anesthesia, cardiopulmonary bypass causing a systemic inflammatory response and oxidative stress that causes pulmonary ischemia-reperfusion injury, type of surgery, pain management, anesthesia protocol, use of blood products, and diaphragmatic dysfunction.

Despite advances in surgical technique and pre- and postoperative care practices in cardiac surgery, PPC is still an important problem. PPC, cost of patient care, increased morbidity and mortality and length of hospital stay elongation. Due to the absence of effective deep inspiration and coughing due to postoperative pain and anxiety, secretion accumulation and gas exchange are ineffective. In a study, it was determined that after coronary artery bypass graft (CABG), 1-20% of patients were hospitalized again in the first 30 days after discharge due to respiratory system complications and 0.4-22.5% of pleural effusion. Various respiratory physiotherapy methods are used for the prevention and treatment of PPC after cardiac surgery. The main purpose of respiratory physiotherapy is to improve ventilation-perfusion compatibility, increase lung volume, increase mucociliary clearance and reduce pain. It has been reported that deep breathing exercises improve postoperative lung expansion and ventilation, resulting in a significant reduction in pulmonary complications. Postoperative respiratory physiotherapy techniques include techniques such as early mobilization, positioning, breathing exercises, active breathing techniques cycle, as well as the use of different mechanical devices such as incentive spirometry (IS), positive expiratory pressure mask therapy, and continuous positive airway pressure. Incentive spirometry (IS) is a mechanical breathing device that provides slow deep breathing and gives visual feedback and is used as one of the important interventions in the prevention of PPC in patients who have been undergoing open heart surgery for many years. Deep breathing exercise training with IS is given to the patients in the preoperative period, and its application is started in the postoperative period. However, it has been reported that insufficiency of physical adaptation and respiratory muscle weakness in the preoperative period are closely related to PPC, which causes prolonged hospital stay and increased mortality. In a meta-analysis study examining the effectiveness of preoperative exercise training for the prevention of PPC in adults undergoing major surgery, it was found that preoperative exercise training minimizes the use of hospital resources, improves physical fitness, and reduces the risk of developing PPC, regardless of the type of surgery. In a meta-analysis study examining the effectiveness of preoperative and postoperative rehabilitation in patients with lung cancer, it was determined that preoperative rehabilitation was effective in reducing postoperative pulmonary complications and hospital stay associated with lung cancer surgery. In studies examining the effectiveness of deep breathing exercise with IS on the development of PPC in cardiac surgery patients, it is seen that IS application is performed in the postoperative period, it is noteworthy that there is no study examining the effectiveness of preoperative IS application.

In the light of this information, the aim of this study is to evaluate the effect of deep breathing exercise with incentive spirometry initiated in the preoperative period on pulmonary function and complications in patients undergoing open heart surgery.

Research Hypotheses H1: Oxygen saturation measured using the pulse oximeter TBY200 will be significantly higher in patients undergoing open heart surgery and initiating deep breathing exercise with IS in the preoperative period.

H2: Arterial blood gas parameters (pH: 7.35-7.45, PaCO2:35-45 mmHg PaO2:80-100 mmHg, SaO2: 95-97%, HCO3:22-26 mEq/L) in patients who underwent open heart surgery and started deep breathing exercise with IS in the preoperative period will have significantly more normal values.

H3: Postoperative pulmonary complications will develop significantly less in patients undergoing open heart surgery and initiating deep breathing exercise with IS in the preoperative period.

H4: In patients undergoing open heart surgery and initiating deep breathing exercise with IS in the preoperative period, the duration of mechanical ventilation will be significantly shorter.

H5: In patients undergoing open heart surgery and initiating deep breathing exercise with IS in the preoperative period, the length of stay in the intensive care unit will be significantly shorter.

H6: In patients undergoing open heart surgery and initiating deep breathing exercise with IS in the preoperative period, the postoperative hospital stay will be significantly shorter.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Able to speak and understand Turkish,
* Conscious, oriented and cooperative,
* First time undergoing cardiac surgery,
* In the Preoperative Chest Diseases Consultation, it was determined that there was no lung pathology and bronchodilator treatment was not started,
* Coronary artery bypass graft (CABG), heart valve surgery or combined open cardiac surgery,
* Having a score of 1 on the Medical Research Council Scale (MRCS),

Exclusion Criteria:

* Emergency surgical intervention applied,
* Complete (100%) occlusion of the left main coronary (LMCA) or right main coronary artery,
* With concomitant vascular aneurysm,
* Chronic respiratory system disease (Asthma, COPD, bronchiectasis, bullous lung, etc.),
* Those who do not agree to participate in the study,
* Died in the process of working,
* Patients for whom data cannot be collected will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Respiratory rate1 | within 24 hours of hospitalization
  the respiratory rate will be counted by the research nurse the first day of hospitalization.
Respiratory rate2 | up to 24 hours before surgery
  the respiratory rate will be counted by the research nurse the day before surgery.
Respiratory rate3 | up to 24 hours
  the respiratory rate will be counted by the research nurse the day after surgery.
Respiratory rate4 | up to 24 hours
  the respiratory rate will be counted by the research nurse on the day of discharge.
SpO2 level1 | within 24 hours of hospitalization
  the SpO2 level of patients will be evaluated the first day of hospitalization.
SpO2 level2 | up to 24 hours
  the SpO2 level of patients will be evaluated the day before surgery.
SpO2 level3 | up to 24 hours
  the SpO2 level of patients will be evaluated the day after surgery.
SpO2 level4 | up to 24 hours
  the SpO2 level of patients will be evaluated on the day of discharge.
Arterial blood gas parameters-pH1 | within 24 hours of hospitalization
  Arterial blood gas parameters of the patients on the first day of hospitalization will be evaluated
Arterial blood gas parameters-O2-1 | within 24 hours of hospitalization
  Arterial blood gas parameters of the patients on the first day of hospitalization will be evaluated
Arterial blood gas parameters-CO2-1 | within 24 hours of hospitalization
  Arterial blood gas parameters of the patients on the first day of hospitalization will be evaluated
Arterial blood gas parameters-saO2-1 | within 24 hours of hospitalization
  Arterial blood gas parameters of the patients on the first day of hospitalization will be evaluated
Arterial blood gas parameters-HCO3-1 | within 24 hours of hospitalization
  Arterial blood gas parameters of the patients on the first day of hospitalization will be evaluated
Arterial blood gas parameters-pH2 | up to 24 hours
  Arterial blood gas parameters of the patients before surgery will be evaluated .
Arterial blood gas parameters-O2-2 | up to 24 hours
  Arterial blood gas parameters of the patients before surgery will be evaluated
Arterial blood gas parameters-CO2-2 | up to 24 hours
  Arterial blood gas parameters of the patients before surgery will be evaluated
Arterial blood gas parameters-saO2-2 | up to 24 hours
  Arterial blood gas parameters of the patients before surgery will be evaluated
Arterial blood gas parameters-HCO3-2 | up to 24 hours
  Arterial blood gas parameters of the patients before surgery will be evaluated
Arterial blood gas parameters-pH-3 | up to 24 hours
  Arterial blood gas parameters of the patients postoperative first day will be evaluated .
Arterial blood gas parameters-pO2-3 | up to 24 hours
  Arterial blood gas parameters of the patients postoperative first day will be evaluated .
Arterial blood gas parameters-pCO2-3 | up to 24 hours
  Arterial blood gas parameters of the patients postoperative first day will be evaluated .
Arterial blood gas parameters-psaO2-3 | up to 24 hours
  Arterial blood gas parameters of the patients postoperative first day will be evaluated .
Arterial blood gas parameters-HCO3 | up to 24 hours
  Arterial blood gas parameters of the patients postoperative first day will be evaluated .
Arterial blood gas parameters-pH.4 | up to 24 hours
  Arterial blood gas parameters of the patients on the day of discharge will be evaluated .
Arterial blood gas parameters-pO2.4 | up to 24 hours
  Arterial blood gas parameters of the patients on the day of discharge will be evaluated .
Arterial blood gas parameters-pCO2.4 | up to 24 hours
  Arterial blood gas parameters of the patients on the day of discharge will be evaluated .
Arterial blood gas parameters-psaO2.4 | up to 24 hours
  Arterial blood gas parameters of the patients on the day of discharge will be evaluated .
Arterial blood gas parameters-HCO3.4 | up to 24 hours
  Arterial blood gas parameters of the patients on the day of discharge will be evaluated .
Posteroanterior chest X-ray-1 | within 24 hours of hospitalization
  All patients' first PA X-rays taken on the first day of hospitalization will be evaluated by the investigator.
Posteroanterior chest X-ray-2 | up to 24 hours
  All patients' last PA X-rays taken on the day of dischargewill be evaluated by the investigator.
Postoperative pulmonary complication | Before discharge (up to 14 days)
  Defined as the occurrence of at least 1 pulmonary complication among atelectasis, pleural effusion, respiratory failure, pneumonia, pneumothorax, bronchospasm, or aspiration pneumonia. The presence of the developing condition, diagnosed by the doctor, was determined as the criterion. This will be evaluated by the Investigator physician and nurse.

SECONDARY OUTCOMES:
Length of stay in mechanical ventilation | up to 24 hours
  The time from the moment the patients are intubated until they are extubated will be recorded in "hours".
Length of stay in intencive care unit(ICU) | Before discharge ICU (up to 1 day)
  The time from the moment the patients are ICU. It will be recorded in "days".
Length of hospitalization | Before discharge (up to 14 days)
  Postoperative stay will be calculated in days from the first postoperative day. This will be evaluated by the investigative nurse. It will be recorded in "days"

CONTACTS AND LOCATIONS:
Overall Officials: Hatice ÖNER CENGİZ, PhD., Study Director — Ankara University; Zeynep ULUŞAN ÖZKAN, MD, Principal Investigator — university of health sciences ankara education and research hospital; Eylem GANİ, Nurse, Principal Investigator — university of health sciences ankara education and research hospital
Locations (1):
- Hatice ÖNER CENGİZ, Altındağ, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oner Cengiz H, Ulusan Ozkan Z, Gani E. The effect of preoperative deep breathing exercise with incentive spirometer initiated in the preoperative period on respiratory parameters and complications in patients underwent open heart surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Jan 24;25(1):36. doi: 10.1186/s12871-025-02902-9. PMID 39856565